CLINICAL TRIAL: NCT00004424
Title: Randomized Study of Propofol Versus Fentanyl and Midazolam in Pediatric Patients Requiring Mechanical Ventilation and Sedation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Case Western Reserve University (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13353; CWRU-FDR000852
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Respiration Disorders
Keywords: disease-related problem/condition; oncologic disorders; pulmonary complications; rare disease; Respiration, Artificial
MeSH Terms: conditions — Respiration Disorders; Rare Diseases; Respiratory Aspiration | interventions — Fentanyl; Midazolam; Propofol

INTERVENTIONS:
Drug: fentanyl
Drug: Midazolam
Drug: propofol

SUMMARY:
OBJECTIVES:

I. Assess the degree of amnesia afforded by study sedatives relative to the patient's intensive care unit experiences.

II. Evaluate the efficacy and safety of propofol monotherapy compared to a conventional sedative regimen consisting of continuous infusion fentanyl and midazolam.

III. Perform a detailed pharmacoeconomic evaluation of propofol sedation compared to combination drug therapy in acutely ill, mechanically ventilated pediatric patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double blind study.

Patients are randomized to receive either a continuous infusion of propofol or a continuous infusion combination of fentanyl and midazolam preceded by a loading dose. Sedative doses may be reduced if necessary. Treatment is continued until sedation is no longer needed, any other sedative therapy is administered, or unacceptable toxicity is experienced.

Patients are assessed after extubation, just prior to hospital discharge, and then every 2 months for 6 months after hospital discharge.

ELIGIBILITY:
* Patients admitted to the Rainbow Babies and Children's Hospital Pediatric Intensive Care Unit who require mechanical ventilation and sedation therapy
* Mean COMFORT score must be greater than 26 after 3 consecutive scores are obtained at 2 minute intervals over 6 minutes
* No other concurrent sedative therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 1996-07; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Michael Deneal Reed, Study Chair — Case Western Reserve University